CLINICAL TRIAL: NCT01057277
Title: BrUOG-H&N-229-RAD001, Cisplatin and Concurrent Radiation for Locally Advanced, Inoperable Head and Neck Cancer: A PHASE I STUDY- Novartis CRAD001CUS134T
Brief Title: RAD001, Cisplatin and Concurrent Radiation for Locally Advanced, Inoperable Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pharmaceutical co- re aligned their specialties- no longer will fund H&N ca
Sponsor: howard safran (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Memorial Hospital of Rhode Island (Other); Roger Williams Medical Center (Other)
Responsible Party: Sponsor-Investigator, howard safran, Principle Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-H&N-229
Record Dates: First submitted 2009-12-09; First posted 2010-01-27 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Advanced Inoperable Head & Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001(Afinitor) (Experimental): Radiation 47 days Cisplatin day 1,8,15,22,29,36,43 RAD001 Day 1 according to assigned group to day 47
  Interventions: Drug: RAD001(Afinitor)

INTERVENTIONS:
Drug: RAD001(Afinitor) — Rad001 in combination withCisplatin and Concurrent RT
  Other Names: Afinitor

SUMMARY:
The purpose of this study is to determine if RAD001, to a maximum dose of 10 mg/day, can be safely administered with cisplatin, and concurrent radiotherapy, for patients with locally advanced, inoperable, squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
To perform a phase I study of RAD001, to a maximum dose of 10 mg/day, with cisplatin, and concurrent radiotherapy, for patients with locally advanced, inoperable, squamous cell carcinoma of the head and neck

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven (from primary lesion and/or lymph nodes) diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx;
* Stage III or IV disease. Patients are unresectable or resection would produce severe impairment or disfiguration.
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:
* History/physical examination within 4 weeks prior to registration
* Chest x-ray (or Chest CT scan or PET/CT scan) within 6 weeks prior to registration.
* CT scan, Pet CT, or MRI of the head and neck (of the primary tumor and neck nodes).
* Zubrod Performance Status 0-1;
* Age > 18;
* Adequate bone marrow function, defined as ANC > 1,500 cells/ul and Platelets > 100,000 cells/ul and Hgb > 9mg/dl.
* Bilirubin < 1.5x upper limit of normal, (For patients with Gilbert's disease as the sole cause of elevated bilirubin, they are eligible if the direct bilirubin is < than 1.5x upper limit of normal)
* AST or ALT < 2.5x the upper limit of normal.
* Adequate renal function, defined as follows:
* Creatinine clearance (CC) ≥ 50 ml/min within 2 weeks prior to registration determined by:

  24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
* INR and PTT < 1.5 x uln. (Anticoagulation is allowed if target INR < 1.5 on a stable dose of warfarin or a stable dose of LMW heparin for > 2 weeks prior to starting treatment.)
* Pregnancy test within 7 days prior to administration of RAD001for women of childbearing potential.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study (until at least 60 days following the last study treatment); If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication and values have been rechecked.
* EKG within 6 weeks of study entry
* Signed informed consent

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3years.
* Patients with simultaneous primaries or bilateral tumors are excluded. Patients with nasopharyngeal cancer and unknown primaries are excluded.
* Gross total excision (e.g., by tonsillectomy) of the primary tumor; however, partial removal of the tumor to alleviate an impending airway obstruction does not make the patient ineligible.
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Initial surgical treatment, excluding diagnostic biopsy of the primary site or nodal sampling of neck disease; radical or modified neck dissection is not permitted.
* Severe, active co-morbidity, defined as follows:
* Current uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure.
* Transmural myocardial infarction within the last 6 months;
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration defined as oxygen saturation that is < 88% at rest on room air.
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
* Any uncontrolled condition, which in the opinion of the investigator, would interfere in the safe and timely completion of study procedures;
* Pregnant or lactating women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception ; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Prior allergic reaction to the study drug(s) involved in this protocol;
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis or serum pregnancy test within 7 days prior to administration of RAD001)
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy etc)
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of the start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring anesthesia) or patients that may require major surgery during the course of the study.
* Prior treatment with any investigational drug within the preceding 4 weeks.
* History of noncompliance to medical regeimens.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Lifespan
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD001(Afinitor)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD001(Afinitor)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 58.6 [49 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Response
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | RAD001(Afinitor)
Number analyzed (Participants) | 3
participants | NA — Study was stopped early and patient's were only assessed for 6 months post drug- no responses seen

ADVERSE EVENTS:
Arm/Group | RAD001(Afinitor)
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001(Afinitor) (N=3)
vomitting (Investigations) | 1 (1)
nausea (Investigations) | 1 (1)
colitis (Investigations) | 1 (1)
acute renal failure (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001(Afinitor) (N=3)
mucositis (Investigations) | 1 (1)
obstructed trach- mucous (Investigations) | 1 (1)
vomitting (Investigations) | 1 (1)
nausea (Investigations) | 2 (2)
diarrhea (Investigations) | 1 (1)
dehydration (Investigations) | 2 (2)
pain-mouth (Investigations) | 1 (1)
wt loss (Investigations) | 2 (2)
fatigue (Investigations) | 2 (2)
edema-face (Investigations) | 1 (1)
tinnitus (Investigations) | 1 (1)
dysphagia (Investigations) | 1 (1)
URI (Investigations) | 1 (1)
wound infection (Investigations) | 1 (1)
neuropathy (Investigations) | 1 (1)
dyspepsia (Investigations) | 1 (1)
SOB (Investigations) | 1 (1)
lymphopenia (Investigations) | 1 (1)
increased creatinine (Investigations) | 1 (1)
increased BUN (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No